CLINICAL TRIAL: NCT04168359
Title: A Clinical Application Study of a CT Guided Small Pulmonary Nodule Puncture and Positioning Device Based on Pre-filled Absorbable Semi-barbed Wire
Brief Title: Semi-barbed Suture for Pulmonary Small Nodules Localization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Aerospace General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: JH.2017.0579
Record Dates: First submitted 2019-11-17; First posted 2019-11-19 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Suture; Nodule, Solitary Pulmonary; Video-Assisted Thoracoscopic Surgery
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Semi-barbed Sutures Localization Group (Experimental): Patients with pulmonary nodules requiring CT-guided puncture positioning before thoracoscopic surgery
  Interventions: Device: absorbable semi-barbed suture

INTERVENTIONS:
Device: absorbable semi-barbed suture — Positioning the intrapulmonary nodules of patient in this group with a absorbable semi-barbed suture positioning device

SUMMARY:
Hookwire and microcoil are currently the most widely used localization instruments. Although their success rate is relatively high in preoperative localization attempts, they may lead to consequences that negatively affect patient outcomes, such as pain because of the metal's hardness, localization failure due to wire detachment, and the presence of permanent traces of metal and foreign bodies .

To overcome these disadvantages, we designed an absorbable semi-barbed suture to localize small intrapulmonary nodules (patent number: ZL201821444387.X).

The results of the previous animal experiments were satisfactory, and it is now necessary to recruit 10 patients for clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. solid nodules with a diameter2cm and distance to visceral pleura 0.5cm；
2. GGN；
3. part-solid GGN, with a solid portion1cm and distance to the visceral pleura 1cm；
4. Patients with nodules at a deep location, who underwent localization to facilitate localization in the resected specimen by a pathologist

Exclusion Criteria:

1. The lesion site is not suitable for percutaneous lung puncture;
2. those who have pneumothorax and pleural effusion;
3. Poor general condition, severe damage to cardiopulmonary function, cachexia, and inability to tolerate surgery;
4. Those who refuse surgery;
5. Those who did not sign the informed consent form.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
Success rate | half an hour after locating
  Successfully located around the small nodules in the lungs, no dislocation occurred

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing aerospace general hospital, Beijing, Beijing Municipality, China